CLINICAL TRIAL: NCT04453306
Title: Treatment of Obesity With Topiramate in Patients With Polycystic Ovary Syndrome: a Double-blind Placebo-controlled Clinical Trial
Brief Title: Treatment of Obesity With Topiramate in Patients With Polycystic Ovary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 140228
Record Dates: First submitted 2020-06-23; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Obesity; Polycystic Ovary Syndrome; Hyperandrogenism
MeSH Terms: conditions — Obesity; Polycystic Ovary Syndrome; Hyperandrogenism | interventions — Topiramate

STUDY DESIGN:
Intervention Model Description: Double-blind Placebo-controlled Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: participants, caregivers, researchers and outcome assessors are blinded to the medications participants are receiving. Participants receive pills with identical size, color and taste between the placebo and the active drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): Patients with the same characteristics as the intervention group. Bottles containing 30 white and green tablets are provided to the participants. The number of bottles is anticipated according to the day of the next appointment. Patients should take 2 tablets bedtime with a full glass of water.
  Bottles are labeled as TPMT100 or TPMT200. The dosage of each tablet is 25 mg, totaling 50 mg / day. The dosage is doubled at 3 months if the patient does not lose at least 3% of the initial weight.
  Interventions: Drug: Placebo
- intervention (Experimental): Patients with the same characteristics as the placebo group. Bottles containing 30 white and green tablets are provided to the participants. The number of bottles is anticipated according to the day of the next appointment. Patients should take 2 tablets bedtime with a full glass of water.
  Bottles are labeled as TPMT100 or TPMT200. The dosage of each tablet is 25 mg, totaling 50 mg / day. The dosage is doubled at 3 months if the patient does not lose at least 3% of the initial weight.
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — topiramate 25mg is coated in tablets in an independent laboratory
  Arms: intervention
Drug: Placebo — innocuous substance is coated in tablets in an independent laboratory
  Arms: placebo

SUMMARY:
Treatment of obesity related to Polycystic Ovary Syndrome with topiramate or placebo to assess improvement of clinical and laboratory parameters after 6 months of follow-up

DETAILED DESCRIPTION:
Randomized double blind placebo-controlled clinical trial. Polycystic ovary syndrome (PCOS) is a frequent endocrinopathy, affecting more than 10% of women of reproductive age. It is associated with a higher prevalence of obesity and insulin resistance, with a higher risk for diabetes, dyslipidemia and hypertension. Topiramate is a drug used in the treatment of epilepsy and migraine prophylaxis since the 1990s and several studies show an association with weight loss. This medicine is administered in combination with phentermine in other countries, with variable weight loss. Despite evidence of the benefit of topiramate for weight loss, there is still no record of studies evaluating this drug in patients with PCOS for the treatment of obesity. The objective of this project is to evaluate the results of treatment with topiramate in terms of weight reduction, reduction of serum androgens and changes in body composition, in patients with PCOS and obese, associated with a low-calorie diet, over a period of six months. Eighty patients with PCOS (18 to 40 years old) seen at the HCPA Endocrinology Service outpatient clinic who are overweight with a BMI> or = 27 kg / m2 associated with at least one comorbidity or obesity (BMI 30-40) will be included. Patients will be randomized to 2 groups: Topiramate and Placebo and the 2 groups will receive a low-calorie diet.

Anthropometric, clinical, hormonal, nutritional and body composition assessment will be performed before, during and after treatments. It is expected to determine whether the addition of topiramate to dietary treatment can improve metabolic, hormonal and weight loss outcomes in women with PCOS.

Research Objective: General objective: To evaluate the results of treatment with topiramate in patients with PCOS and obese, associated with a low-calorie diet, in six months of treatment.

Specific objectives: To evaluate the response to the proposed treatment in terms of weight reduction and body mass index (BMI), reduction of serum androgens, changes in body composition, in addition to assessing minor psychiatric disorders possibly associated through the Self-Reporting screening questionnaire. Questionnaire (SRQ-20).

Assessment of Risks and Benefits: The risks of the project are mainly related to the use of the drug topiramate. This drug has an extensive list of adverse effects, in addition to the side effect on appetite and weight, the most common are paresthesias, drowsiness, lethargy, attention disorder, mood disorders, depression, taste changes and psychomotor disorders. However, studies show that the majority of adverse reactions were mild to moderate in severity. Other risks inherent to the study are the absence of previous studies in the target population and discomfort in relation to the number of visits, additional tests and blood samples for an extended period of 6 months. The benefits of the study are related to the acquisition of knowledge and the likely positive results may benefit future patients.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 40 years
* diagnostic criteria for PCOS
* overweight with a BMI ≥ 27 kg / m² associated with at least one comorbidity (hypertension, type 2 diabetes mellitus, dyslipidemia) or obesity with a BMI between 30 and 45 kg / m² with or without comorbidities

Exclusion Criteria:

* severe systemic arterial hypertension (≥180 / 100 mmHg)
* pregnant or lactating women
* diabetics using sulfonylurea or insulin
* any known allergy or intolerance to topiramate medication

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change of Body Mass index (BMi) at 6 months | 6 months
  change of Body Mass index (BMi) in kg/m² from the baseline; weight and height will be combined to report BMI
change in the modified Ferriman-Gallwey Hirsutism Score (mFG) at 6 months | 6 months
  In the modified method, hair growth is rated from 0 (no growth of terminal hair) to 4 (extensive hair growth) in each of the nine locations (Upper lip, Chin, Chest, Upper back, Lower back, Upper abdomen, Lower abdomen, Upper arms, Thighs). A patient's score may therefore range from a minimum score of 0 to a maximum score of 36. A score of 6 or higher will be adopted as indicative of androgen excess.
Change of testosterone at 6 months | 6 months
  Change of testosterone (ng/mL) at 6 months from the baseline
Change of glucose at 6 months | 6 months
  Change of glucose(mg/dL) at 6 months from the baseline
Change of triglyceride at 6 months | 6 months
  Change of triglyceride (mg/dL) at 6 months from the baseline
Change of High-density lipoprotein (HDL) at 6 months | 6 months
  Change of HDL cholesterol (mg/dL) at 6 months from the baseline
Change of total cholesterol at 6 months | 6 months
  Change of total cholesterol (mg/dL) at 6 months from the baseline
Change of Low-density lipoprotein (LDL) at 6 months | 6 months
  Change of LDL cholesterol (mg/dL) at 6 months from the baseline. LDL cholesterol will be calculated with the Friedewald formula, an estimation of LDL-c level that uses the following levels of total cholesterol (TC), triglycerides (TG), and high-density lipoprotein cholesterol (HDL-c): LDL-c (mg/dL) = TC (mg/dL) - HDL-c (mg/dL) - TG (mg/dL)/5
Change of homeostatic model assessment (HOMA-IR) at 6 months | 6 months
  Change of HOMA-IR at 6 months from the baseline. HOMA-IR will be calculated according to the formula: fasting insulin (µU/L) x fasting glucose (nmol/L)/22.5.
change in systolic blood pressure at 6 months | 6 months
  change in systolic blood pressure (mmHg) at 6 months from baseline.
change in diastolic blood pressure at 6 months | 6 months
  change in diastolic blood pressure (mmHg) at 6 months from baseline.

SECONDARY OUTCOMES:
change of body composition at 6 months | 6 months
  Change in body composition evaluated through Dual-energy X-ray absorptiometry (DXA) from the baseline
Change in anxiety score at 6 months | 6 months
  Change in anxiety score, assessed through the self-report questionnaire-20 (SRQ 20), consisting of 20 questions with a yes / no answer, assigning 1 point to the "yes" answer. A cut-off point of 8 or more indicates an anxiety disorder, with a minimum of zero and a maximum of 20 points.

CONTACTS AND LOCATIONS:
Overall Officials: Poli Mara Spritzer, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided